CLINICAL TRIAL: NCT00179426
Title: Antiseizure Medication-Induced Elevation of Serum Estradiol and Reproductive Dysfunction in Men With Epilepsy
Brief Title: Effect of Antiseizure Medication on Hormone Levels and Sexual Function in Men With Epilepsy
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Andrew Herzog, Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2001P000596
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Seizure Disorder; Epilepsy
Keywords: Seizure Disorder; Hypogonadism; Sexual Function; Epilepsy
MeSH Terms: conditions — Epilepsy; Hypogonadism

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of this study is to determine if antiseizure drugs affect hormone levels and sexual function in men with seizures.

DETAILED DESCRIPTION:
This study involves donating two small tubes of blood for hormonal testing, which will be drawn at the same time as your routine blood draw for the monitoring of your antiseizure medication. You will also be asked to fill out a short confidential questionnaire regarding your sexual interest and function.

ELIGIBILITY:
Inclusion Criteria:

* Must be a male between 18-50 years of age
* Must have seizures
* Must be on antiseizure medication for at least six months duration

Exclusion Criteria:

* Must not have taken hormones, major tranquilizers or antidepressants for at least 3 months

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175
Dates: Start 1999-10; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G. Herzog, M.D., M.Sc., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Herzog AG, Drislane FW, Schomer DL, Pennell PB, Bromfield EB, Kelly KM, Farina EL, Frye CA. Differential effects of antiepileptic drugs on sexual function and reproductive hormones in men with epilepsy: interim analysis of a comparison between lamotrigine and enzyme-inducing antiepileptic drugs. Epilepsia. 2004 Jul;45(7):764-8. doi: 10.1111/j.0013-9580.2004.60703.x. PMID 15230699